CLINICAL TRIAL: NCT06535321
Title: Effects of Vibration Training Combined With Kinesio Taping on Delayed Onset Muscle Soreness of Athletes' Knee Joints: A Randomised Controlled Trial
Brief Title: Delayed Onset Muscle Soreness of Athletes
Acronym: DOMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Sport University (Other)
Responsible Party: Principal Investigator, Cheng Liang, Director, Chengdu Sport University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: No: 2103; 2024NSFSC0681 (Other Grant/Funding Number: Natural Science Foundation of Sichuan Province)
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: Delayed Onset Muscle Soreness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): After modelling, when the vibration platform is closed, all participants of the control group completed the same action as vibration training.
  Interventions: Other: vibration training
- Vibration group (Experimental): For the vibration group, vibration training was performed immediately after DOMS modelling.
  Interventions: Other: vibration training
- Kinesio group (Experimental): For the kinesio group, Y-shaped kinesio taping was performed 30 min before DOMS modelling.
  Interventions: Other: Y-shaped kinesio taping
- Combined group (Experimental): For the combined group, the vibration group and kinesio group interventions were performed simultaneously.
  Interventions: Other: vibration training; Other: Y-shaped kinesio taping; Other: Combined vibration training and Y-shaped kinesio taping

INTERVENTIONS:
Other: vibration training — After modelling, when the vibration platform is closed, all participants of the control group completed the same action as vibration training.
  Arms: Control
Other: vibration training — For the vibration group, vibration training was performed immediately after DOMS modelling.
  Arms: Combined group; Vibration group
Other: Y-shaped kinesio taping — For the kinesio group, Y-shaped kinesio taping was performed 30 min before DOMS modelling.
  Arms: Combined group; Kinesio group
Other: Combined vibration training and Y-shaped kinesio taping — For the combined group, the vibration group and kinesio group interventions were performed simultaneously.
  Arms: Combined group

SUMMARY:
Study Design:

This study was approved by the Human Experiment Ethics Committee of Chengdu Sport University (No: 2103).

Based on previous research data, G-power software was used to calculate that at least 40 samples were needed.

Participants:

A total of 45 track and field athletes from Sichuan Province, China, were recruited during the off-season in 2024. They were randomly assigned to the vibration group, kinesio taping group, combined group, and control group.

All participants signed informed consent forms and adhered to the Declaration of Helsinki.

DOMS Modeling:

Following previous research, a delayed onset muscle soreness (DOMS) model for athletes' knee joints was established through downhill running.

Detailed oxygen uptake tests were conducted on all participants one week before DOMS modeling, and records were made one week after DOMS modeling.

Intervention Measures:

The vibration group received vibration training immediately after DOMS modeling.

The kinesio taping group had Y-shaped kinesio taping applied 30 minutes before DOMS modeling.

The combined group received both vibration training and kinesio taping simultaneously.

Assessment Methods:

The degree of pain at the DOMS site for participants was evaluated using a Visual Analogue Scale (VAS).

The concentration of creatine kinase (CK) in the serum of participants was detected using an RT-9600 automatic biochemical analyzer, and serum interleukin-6 (IL-6) was detected by enzyme-linked immunosorbent assay (ELISA).

An IsoMed 2000 isokinetic tester was used to perform a 60°/s extension test on the participants' knees.

Data Collection:

VAS scores, serum CK and IL-6 levels, and peak torque of knee extension were collected at different time points before and after DOMS modeling.

DETAILED DESCRIPTION:
Materials and Methods Participants This study was approved by the Human Experiment Ethics Committee of Chengdu Sport University (No: 2103). We referred to our previous research on the effect of vibration training on DOMS in athletes1 and the research on the effect of kinesio taping on DOMS in athletes. Considering the experimental design of four groups and five measurements per group, about 5% of the samples were lost. The VAS scores, IL-6 levels and CK levels as indicators of DOMS exhibited high sensitivity and specificity. Using G-power software, the effect size of 0.3 was selected.1,12,14 Power was set at 0.8, and the significance level was set at 0.05. At least 40 samples were needed for calculation.

Track and field athletes from Sichuan Province, China, were recruited during the off-season in 2024. Eligibility criteria were as follows: athletes who performed regular training, ranked in the top 3 in a provincial competition and trained at least 5days per week, with a minimum of 4 h each day. This training encompassed, but was not limited to, strength training, endurance training, skill drills and competitive preparation. The study was in line with the Declaration of Helsinki, and the participants were aware of the study intention and signed informed consent. Exclusion criteria were as follows: lower limb joint injury and systematic exercise training in the last week. A total of 45 participants (male/female: 26/19) meeting the criteria were recruited, and no sample loss was observed throughout the experimental process. The participants were divided into the vibration group (n = 11), kinesio group (n =11), combined group (vibration training + kinesio taping, n = 12) and control group (n = 11) by digital random grouping. No statistically in age, height and body mass amongst groups were observed.

DOMS Modelling Referring to our previous experimental design for DOMS modelling of athletes' knee joints,1 we performed a detailed oxygen uptake test (Cortex Cardiopulmonary Function Test System, Model: Metalyzer 3B, Germany) on all participants at 1 week before DOMS modelling. A detailed record was made 1 week after DOMS modelling. Participants performed downhill running on a treadmill (ICON, Model: NETL28717, USA; gradient of -10°, 5 groups, 8 min/group, 2 min of flat walking between groups). According to the maximum oxygen uptake, exercise intensity was matched for each participant, ensuring that all participants included had similar aerobic capacity and could maintain similar intensity during downhill running to complete DOMS modelling. Participants wore a Polar watch (Finland, Model: M430) throughout the course to monitor their heart rate, ensuring that 80% of maximum heart rate was maintained during downhill running. If the heart rate was too low or too high, the treadmill speed was adjusted appropriately. Within 72 h after DOMS modelling, we followed up with the participants to ensure that they did not undergo other training activities or treatments. Pain is a significant indicator of DOMS. In this study, the success of DOMS modelling was determined by comparing the VAS scores of participants immediately after modelling with the baseline scores. We observed that the average VAS scores for knee joint pain increased from 0.11 (0.01-0.21) to 2.21 (0.54-3.53) amongst all participants. Thus, the participants experienced varying degrees of DOMS.

The following interventions were performed on each group in this study. For the vibration group, vibration training was performed immediately after DOMS modelling. For the kinesio group, Y-shaped kinesio taping was performed 30 min before DOMS modelling. After modelling, when the vibration platform is closed, all participants of the kinesio group and control group completed the same action as vibration training. For the combined group, the vibration group and kinesio group interventions were performed simultaneously.

Vibration Training On the basis of our previous experimental design and research results of vibration training intervention for athletes, a vibration training intervention with a frequency of 50 Hz, an amplitude of 3 mm and a duration of 10 min was selected.1 Using a Power Plate vibrating platform (Model: Power Plate pro5TM, USA), vibration training was performed on the participants of the vibration group and combined group who had completed DOMS modelling under the guidance of the experimenter. The participants performed a half squat (3 min) and a lunge pull (3.5 min on each side) on the vibrating platform.1 The kinesio group and control group participants performed the same number of sets and times as the vibration group and combined group participants when the vibrator was turned off. Vibration training was performed only once, immediately after DOMS molding.

Kinesio Taping Y-shaped kinesio taping was performed 30 min before DOMS modelling.14 The participants took a sitting position, keeping their knees bent at 90°. Professional physiotherapists used 5 cm × 5 m intramuscular adhesive tape (LP Support, USA, size: 5 cm × 5 m, colour: blue) to tape the bilateral vastus medialis, vastus lateralis and rectus femoris in a 'Y' shape (stretched to 125% of the original length).16 To avoid the detachment of the muscle tape, we re-taped the same operation at 24, 48 and 72 h. During DOMS modelling, most of the participants did not lose the muscle tape, but some participants lost part of the tape, which was re-taped immediately.

This study evaluated the VAS scores, serum CK and IL-6 levels and peak torque of knee extension (60 °/s) before DOMS modelling (baseline and at 24 h before DOMS modelling) and after vibration training (immediately), 24 h, 48 h and 72 h of the participants in the four groups.

VAS Testing The pain degree of the participants at the DOMS site was evaluated by VAS. The participants were asked to draw a vertical line on a 10 cm straight line (0 cm was painless, and 10 cm was the most painful, scored 0-10. The left and right knee joints were drawn once each, and the mean was processed.

Serum IL-6 and CK Testing Our previous methods provide further details.1 About 3 mL of venous blood was collected from the participants, and the CK concentration of the participants at five time points was detected by using an RT-9600 automatic biochemical analyser (kit provided by Shanghai Lanxing Biotechnology Co., Ltd.). Serum IL-6 was detected by enzyme-linked immunosorbent assay (kit provided by Shanghai Varan Biotechnology Co., Ltd.).

Isokinetic Knee Testing An IsoMed 2000 isokinetic tester from Germany was used to perform 60°/s (three times) extension test on the participants' knee. The participants were in a sitting position, and the trunk and hip joints were fixed with a wide binding. The knee joint extension mode was selected with the joint activity of 80°, and the analytical index was peak torque; the test data were averaged on the left and right sides.

ELIGIBILITY:
Inclusion Criteria:

* Athletes who performed regular training, ranked in the top 3 in a provincial competition and trained at least 5days per week, with a minimum of 4 h each day.
* This training encompassed, but was not limited to, strength training, endurance training, skill drills and competitive preparation.
* This study was in line with the Declaration of Helsinki, and the participants were aware of the study intention and signed informed consent.

Exclusion Criteria:

* Lower limb joint injury and systematic exercise training in the last week.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
VAS Testing | 7 Days
  The pain degree of the participants at the DOMS site was evaluated by VAS. The participants were asked to draw a vertical line on a 10 cm straight line (0 cm was painless, and 10 cm was the most painful, scored 0-10. The left and right knee joints were drawn once each, and the mean was processed.
Serum IL-6 Testing | 7 Days
  About 3 mL of venous blood was collected from the participants, and the CK concentration of the participants at five time points was detected by using an RT-9600 automatic biochemical analyser (kit provided by Shanghai Lanxing Biotechnology Co., Ltd.).
CK Testing | 7 Days
  About 3 mL of venous blood was collected from the participants. Serum IL-6 was detected by enzyme-linked immunosorbent assay (kit provided by Shanghai Varan Biotechnology Co., Ltd.).
Isokinetic Knee Testing | 7 Days
  An IsoMed 2000 isokinetic tester from Germany was used to perform 60°/s (three times) extension test on the participants' knee. The participants were in a sitting position, and the trunk and hip joints were fixed with a wide binding. The knee joint extension mode was selected with the joint activity of 80°, and the analytical index was peak torque; the test data were averaged on the left and right sides.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Cheng, Dr, Principal Investigator — Chengdu Sport University

IPD SHARING:
Plan to Share IPD: No